CLINICAL TRIAL: NCT00338676
Title: Aortic Stenosis in Elderly : Determinant of Progression. COFRASA (French Cohort)
Brief Title: Aortic Stenosis in Elderly : Determinant of Progression
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM05003 - P051042
Record Dates: First submitted 2006-06-19; First posted 2006-06-20 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2016-02

CONDITIONS: Aortic Stenosis; Elderly Gravida
Keywords: Aortic stenosis; Elderly
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Aortic stenosis (AS) is AS is caused by calcium deposits in the aortic valve. Calcification is progressive and eventually leads to reduced leaflet motion with obstruction of the left ventricular outflow. The only treatment is surgery. There are evidences that AS is a regulated process with similarities to atherosclerosis but determinants of AS progression are unknown. The study aims at evaluating these determinants and more specifically the role of lipids, inflammation and platelet aggregation.

DETAILED DESCRIPTION:
Aortic stenosis (AS) is the most common valvular disease and the second most common indication for cardiac surgery in Western countries. AS prevalence increases with age and with aging of the population, AS is a major public health problem. AS is due to calcium deposits within the aortic valve. Calcium deposit is progressive and eventually leads to reduced leaflet motion with obstruction of the left ventricular outflow. There is currently no effective medical therapy. Once the stenosis is severe and patients symptomatic, outcome is poor unless surgery (aortic valve replacement) is promptly performed. AS has long been considered as a passive and degenerative process. Recent data challenged this concept, showing that AS is an active and highly regulated process with some similarities to atherosclerosis. However, AS progression is highly variable from one individual to another and determinants of AS progression are poorly known. Their identification is crucial if we want to develop new medical strategies. The aims of the present study are to identify the determinants of AS progression and more specifically to evaluate the role of lipids, inflammation and platelet aggregation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* AS with mean transmitral gradient > 10 mm Hg and aortic valve area < 2 cm2
* No surgical indication

Exclusion Criteria:

* Rheumatic or congenital AS
* Associated valvular disease grade ≥ 2/4
* Indication for surgery (severe AS (aortic valve area < 1 cm2 or < 0.6 cm2/m2 of body surface area and symptoms or congestive heart failure or left ventricular ejection fraction < 50%)
* Renal insufficiency (creatinine clearance < 30 ml /min)
* Left ventricular outflow tract obstruction

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients diagnosed with an at least mild aortic stenosis with no indication for surgery
Sampling Method: Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2006-11; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Progression of aortic stenosis | 2006 - 2017

SECONDARY OUTCOMES:
AS related events | 2006 - 2017

CONTACTS AND LOCATIONS:
Overall Officials: David Messika-Zeitoun, MD, Principal Investigator — Assistance Publique des Hopitaux de Paris
Locations (1):
- Hopital Bichat, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perrot N, Theriault S, Dina C, Chen HY, Boekholdt SM, Rigade S, Despres AA, Poulin A, Capoulade R, Le Tourneau T, Messika-Zeitoun D, Trottier M, Tessier M, Guimond J, Nadeau M, Engert JC, Khaw KT, Wareham NJ, Dweck MR, Mathieu P, Pibarot P, Schott JJ, Thanassoulis G, Clavel MA, Bosse Y, Arsenault BJ. Genetic Variation in LPA, Calcific Aortic Valve Stenosis in Patients Undergoing Cardiac Surgery, and Familial Risk of Aortic Valve Microcalcification. JAMA Cardiol. 2019 Jul 1;4(7):620-627. doi: 10.1001/jamacardio.2019.1581. PMID 31141105
- [Derived] Pawade T, Clavel MA, Tribouilloy C, Dreyfus J, Mathieu T, Tastet L, Renard C, Gun M, Jenkins WSA, Macron L, Sechrist JW, Lacomis JM, Nguyen V, Galian Gay L, Cuellar Calabria H, Ntalas I, Cartlidge TRG, Prendergast B, Rajani R, Evangelista A, Cavalcante JL, Newby DE, Pibarot P, Messika Zeitoun D, Dweck MR. Computed Tomography Aortic Valve Calcium Scoring in Patients With Aortic Stenosis. Circ Cardiovasc Imaging. 2018 Mar;11(3):e007146. doi: 10.1161/CIRCIMAGING.117.007146. PMID 29555836
- [Derived] Arangalage D, Nguyen V, Robert T, Melissopoulou M, Mathieu T, Estellat C, Codogno I, Huart V, Duval X, Cimadevilla C, Vahanian A, Dehoux M, Messika-Zeitoun D. Determinants and prognostic value of Galectin-3 in patients with aortic valve stenosis. Heart. 2016 Jun 1;102(11):862-8. doi: 10.1136/heartjnl-2015-308873. Epub 2016 Feb 19. PMID 26896466
- [Derived] Chin CW, Messika-Zeitoun D, Shah AS, Lefevre G, Bailleul S, Yeung EN, Koo M, Mirsadraee S, Mathieu T, Semple SI, Mills NL, Vahanian A, Newby DE, Dweck MR. A clinical risk score of myocardial fibrosis predicts adverse outcomes in aortic stenosis. Eur Heart J. 2016 Feb 21;37(8):713-23. doi: 10.1093/eurheartj/ehv525. Epub 2015 Oct 21. PMID 26491110
- [Derived] Nguyen V, Cimadevilla C, Estellat C, Codogno I, Huart V, Benessiano J, Duval X, Pibarot P, Clavel MA, Enriquez-Sarano M, Vahanian A, Messika-Zeitoun D. Haemodynamic and anatomic progression of aortic stenosis. Heart. 2015 Jun;101(12):943-7. doi: 10.1136/heartjnl-2014-307154. Epub 2015 Feb 5. PMID 25655063
- [Derived] Cimadevilla C, Cueff C, Hekimian G, Dehoux M, Lepage L, Iung B, Duval X, Huart V, Tubach F, Vahanian A, Messika-Zeitoun D. Prognostic value of B-type natriuretic peptide in elderly patients with aortic valve stenosis: the COFRASA-GENERAC study. Heart. 2013 Apr;99(7):461-7. doi: 10.1136/heartjnl-2012-303284. Epub 2013 Jan 24. PMID 23349346
- [Derived] Hekimian G, Boutten A, Flamant M, Duval X, Dehoux M, Benessiano J, Huart V, Dupre T, Berjeb N, Tubach F, Iung B, Vahanian A, Messika-Zeitoun D. Progression of aortic valve stenosis is associated with bone remodelling and secondary hyperparathyroidism in elderly patients--the COFRASA study. Eur Heart J. 2013 Jul;34(25):1915-22. doi: 10.1093/eurheartj/ehs450. Epub 2013 Jan 17. PMID 23329150